CLINICAL TRIAL: NCT03525691
Title: Enhanced Lung Protective Ventilation With Extracorporeal CO2 Removal During Acute Respiratory Distress Syndrome
Brief Title: Enhanced Lung Protective Ventilation With ECCO2R During ARDS
Acronym: PROVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Principal Investigator, Jerome Allardet-Servent, MD, Principal Investigator, Hôpital Européen Marseille
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-A03647-46
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: ARDS, Human; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Minimal distension (Experimental): Tidal volume 4 ml/kg PBW and positive end-expiratory pressure (PEEP) based on the ARDSNet PEEP/FiO2 table (ARMA) + ECCO2R (sweep gas = 8 L/min, blood flow = 400 mL/min)
  Interventions: Device: Low flow Extracorporeal CO2 removal
- Maximal recruitment (Experimental): Tidal volume 4 ml/kg PBW and PEEP adjusted to maintain a plateau pressure between 23 - 25 cmH2O + ECCO2R (sweep gas = 8 L/min, blood flow = 400 mL/min)
  Interventions: Device: Low flow Extracorporeal CO2 removal
- Standard (Active Comparator): Tidal volume 6 ml/kg PBW and positive end-expiratory pressure (PEEP) based on the ARDSNet PEEP/FiO2 table (ARMA) without ECCO2R (no sweep gas flow, blood flow = 400 mL/min)
  Interventions: Device: Low flow Extracorporeal CO2 removal

INTERVENTIONS:
Device: Low flow Extracorporeal CO2 removal — Low flow Extracorporeal CO2 removal using a 0.67 m² membrane oxygenator (Lilliput 2) and a specific circuit (HP-X) mounted on a RRT monitor (PrismafleX)

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is associated with a mortality rate of 30 - 45 % and required invasive mechanical ventilation (MV) in almost 85 % of patients[1]. During controlled MV, driving pressure (i.e., the difference between end-inspiratory and end-expiratory airway pressure) depends of both tidal volume and respiratory system compliance. Either excessive tidal volume or reduced lung aeration may increase the driving pressure. ARDS patients receiving tidal volume of 6 ml/kg predicted body weight (PBW) and having a day-1 driving pressure ≥ 14 cmH2O have an increased risk of death in the hospital[2]. Seemly, in the LUNG SAFE observational cohort, ARDS patients having a day-1 driving pressure < 11 cmH2O had the lowest risk of death in the hospital[1]. Hence, driving pressure acts as a major contributor of mortality in ARDS, and probably reflects excessive regional lung distension resulting in pro-inflammatory and fibrotic biological processes. Whether decreasing the driving pressure by an intervention change mortality remains an hypothesis; but one of means is to decrease the tidal volume from 6 to 4 ml/ kg predicted body weight (PBW). However, this strategy promotes hypercarbia, at constant respiratory rate, by decreasing the alveolar ventilation. In this setting, implementing an extracorporeal CO2 removal (ECCO2R) therapy prevents from hypercarbia. A number of low-flow ECCO2R devices are now available and some of those use renal replacement therapy (RRT) platform. The investigators previously reported that combining a membrane oxygenator (0.65 m²) within a hemofiltration circuit provides efficacious low flow ECCO2R and blood purification in patients presenting with both ARDS and Acute Kidney injury[3].

This study aims to investigate the efficacy of an original ECCO2R system combining a 0.67 m² membrane oxygenator (Lilliput 2, SORIN) inserted within a specific circuit (HP-X, BAXTER) and mounted on a RRT monitor (PrismafleX, BAXTER). Such a therapy only aims to provide decarboxylation but not blood purification and has the huge advantage to be potentially implemented in most ICUs without requiring a specific ECCO2R device. The study will consist in three periods:

* The first period will address the efficacy of this original ECCO2R system at tidal volume of 6 and 4 ml/kg PBW using an off-on-off design.
* The second part will investigate the effect of varying the sweep gas flow (0-2-4-6-8-10 l/min) and the mixture of the sweep gas (Air/O2) on the CO2 removal rate.
* The third part will compare three ventilatory strategies applied in a crossover design:

  1. Minimal distension: Tidal volume 4 ml/kg PBW and positive end-expiratory pressure (PEEP) based on the ARDSNet PEEP/FiO2 table (ARMA).
  2. Maximal recruitment: 4 ml/kg PBW and PEEP adjusted to maintain a plateau pressure between 23 - 25 cmH2O.
  3. Standard: Tidal volume 6 ml/kg and PEEP based on the ARDSNet PEEP/FiO2 table (ARMA).

ELIGIBILITY:
Inclusion Criteria:

* ARDS moderate or severe (Berlin criteria)
* Onset < 48 h
* Driving pressure ≥ 11 cmH2O

Exclusion Criteria:

* Lack of consent or social protection
* Chronic respiratory failure (requiring Oxygen or NIPPV)
* Severe hypoxemia: PaO2/FIO2 < 80 with PEEP ≥ 18 cmH2O AND FIO2= 1
* Acute Renal Failure requiring RRT
* DNR order or death expected within the next 72 hours
* Planned surgery or transport out-of-ICU expected within the next 72 hours
* Heparin allergy
* Contraindication to jugular vein catheterization
* Intracranial Hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change in PaCO2 | 15 minutes after initiation of ECCO2R at tidal volume of 4 ml/kg PBW.
  20 % decrease in PaCO2 after initiation of ECCO2R at tidal volume of 4 ml/kg PBW (as compared to 4 ml/kg without ECCO2R)

SECONDARY OUTCOMES:
PaCO2 | each 15 minutes up to the third hour (Part I and II of the study). In the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Arterial blood gas analyser (RAPIDPoint 500)
CO2 removal rate | each 15 minutes up to the third hour (Part I and II of the study). In the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using measurements from both the blood side and the gas side (two methods)
Transpulmonary pressure and work of breathing | each 15 minutes up to the third hour (Part I and II of the study). In the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using an oesophageal balloon catheter (NutriVent catheter) and a dedicated monitor (FluxMed, MBMed)
Regional tidal ventilation | each 15 minutes up to the third hour (Part I and II of the study). In the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using an Electrical Impedance Tomography device (BB², Swisstom)
End-expiratory Lung Volume | each 15 minutes up to the third hour (Part I and II of the study). In the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using the nitrogen wash-in wash-out method (Engstrom GE)
Plasma Cytokines | Only in the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using Elisa custom kit (Qiagen) from plasma samples
Pulmonary Cytokines | Only in the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using Elisa custom kit (Qiagen) from BAL samples
Type III Procollagen | Only in the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using both RIA and Elisa methods from plasma and BAL samples
Pulmonary Inflammatory and Fibrotic pathway | Only in the third part, measurement at baseline and at 1 hour and at 22 hours into each arm.
  Using mRNA custom kit RT-PCR analysis (Qiagen) from BAL samples

OTHER OUTCOMES:
Plasma Free Hemoglobin | every 24 hours, up to 72 hours.
  serum samples
Haptoglobin | every 24 hours, up to 72 hours.
  serum samples
Lacticodéshydrogenase (LDH) | every 24 hours, up to 72 hours.
  serum samples
schizocytes | every 24 hours, up to 72 hours.
  serum samples
Bilirubin | every 24 hours, up to 72 hours.
  serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme ALLARDET-SERVENT, MD, Principal Investigator — Hopital Européen Marseille
Locations (1):
- Service de REANIMATION, HOPITAL EUROPEEN MARSEILLE, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Allardet-Servent J, Castanier M, Signouret T, Soundaravelou R, Lepidi A, Seghboyan JM. Safety and Efficacy of Combined Extracorporeal CO2 Removal and Renal Replacement Therapy in Patients With Acute Respiratory Distress Syndrome and Acute Kidney Injury: The Pulmonary and Renal Support in Acute Respiratory Distress Syndrome Study. Crit Care Med. 2015 Dec;43(12):2570-81. doi: 10.1097/CCM.0000000000001296. PMID 26488219